CLINICAL TRIAL: NCT02361866
Title: Randomized, Double Blind, Multicenter, Phase III Study to Evaluate the Effectiveness(Immunogeneicity) and Safety of 'GC1107' Administered Intramuscularly in Healthy Adults
Brief Title: To Evaluate the Effectiveness(Immunogeneicity) and Safety of 'GC1107' Administered Intramuscularly in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GC1107_AD_P3
Record Dates: First submitted 2014-04-22; First posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GC1107 (Experimental): 0.5ml, intramuscular, a single dosing
  Interventions: Biological: GC1107
- Tetanus and Diphtheria(Td vaccine) (Active Comparator): 0.5ml, intramuscular, a single dosing
  Interventions: Biological: Tetanus and Diphtheria(Td vaccine)

INTERVENTIONS:
Biological: GC1107 — 0.5 ml, Intramuscular, single dose(day0)
  Arms: GC1107
Biological: Tetanus and Diphtheria(Td vaccine) — 0.5ml, Intramuscular, single dose(day0) only applicable step1
  Arms: Tetanus and Diphtheria(Td vaccine)

SUMMARY:
The purpose of this study is to evaluate the effectiveness(immunogeneicity) and safety of 'GC1107' administered intramuscularly in healthy Adults.

DETAILED DESCRIPTION:
Randomized, double blind, multicenter, phaseⅢ study

ELIGIBILITY:
Inclusion Criteria:

* healthy Korean adults (age: over 18 years)
* who got the basic vaccination of DTP(Diphtheria, tetanus, pertussis) in the past
* Subjects willing to provide written informed consent and able to comply with the requirements for the study

Exclusion Criteria:

* subjects who have already got the additional vaccination of Td within 5 years
* subjects with antitoxin of diphtheria and tetanus ≥1.0 IU/mL (ELISA)

  * only applicable in step I
* subjects who have not recovered from the acute disease within 2 weeks
* subjects who have the medical history of allergic disease related to the components of investigational drug
* who got the treatment of blood product and immunoglobulin product within 3 months
* females who are pregnant
* females who are breastfeeding
* subjects who are infected from the diphtheria and tetanus
* subjects who have experienced the severe adverse events for the diphtheria and tetanus vaccination
* Subjects who are scheduled to participate in other clinical trial studies during the study
* Subjects who have participated in any other clinical trials within 4 weeks of the administration of the study
* Those who take the other medicine that affects this study or are vaccinated other vaccines
* Subject who have received adrenocortical hormones or immunosuppressive drug within 4weeks of enrollment
* Subjects with a history of chronic disease obstacles to the study.
* Subjects who have episode of acute febrile (at least 37.4) after injection of vaccine during the study
* Subject who have plan of operation during the study.
* Individuals with other clinically significant medical or psychological condition who are considered by the investigator to be ineligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
seroprotection rate of diphtheria and tetanus | 28days

SECONDARY OUTCOMES:
GMT (Geometric Mean Titer) | 28days
Boosting response of diphtheria and tetanus compared participants with before and after the injection | 28days
  Boosting response is defined as more 4 times increase of the antibody titer after the injection
solicited adverse events | 7days
unsolicited adverse events | 28 days
Seroprotection rate according to the respective age group | 28days
GMT according to the respective age group | 28days

CONTACTS AND LOCATIONS:
Overall Officials: JungHyeon Choi, MD, Principal Investigator — Incheon St. Mary's Hospital Catholic University
Locations (1):
- Incheon St. Mary's Hospital Catholic Univ., Incheon, Bupyeong 6-dong, Bupyeong-gu,, South Korea

REFERENCES:
- [Derived] Lee J, Choi JH, Wie SH, Park SH, Choi SM, Lee MS, Kim TH, Lee HJ, Kang JH. A Phase III Study to Evaluate the Immunogenicity and Safety of GC1107 (Adult Tetanus Diphtheria Vaccine) in Healthy Adults. J Korean Med Sci. 2019 Jan 16;34(4):e31. doi: 10.3346/jkms.2019.34.e31. eCollection 2019 Jan 28. PMID 30686952